CLINICAL TRIAL: NCT00678756
Title: Investigation of Antipsoriatic Effects of UVB-induced Synthesis of 1alpha, 25-Dihydroxyvitamin D3 (1alpha, 25(OH)2D3, Calcitriol)in Keratinocytes of Psoriatic Skin, Using Cytochrom-P(CYP)Inhibitor Ketokonazol
Acronym: VITAKET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. med. Gottfried Wozel, Technical University Dresden, Department of Dermatology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-VITAKET
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis vulgaris,; vitamin D, UVB-phototherapy, ketokonazol,; Optical Coherence Tomography,; local PASI, Nizoral
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ketokonazol 2% cream — twice a day at 2 times,2 out of 5 areas have to be treated for 4 weeks/7 days a week
  Other Names: Nizoral cream
Radiation: UVB-radiation 311nm — 3 out of 5 areas are radiated for 4 weeks every MO/DI/DO/FR starting MED orientated, intensified everytime 0,03 J/qcm
  Other Names: UVB Radiation, phototherapy, narrow-band ultraviolet B phototherapy

SUMMARY:
Exploration of antipsoriatic effects of UVB-therapy +/- CYP-inhibitor Ketokonazol on affected psoriatic skin

ELIGIBILITY:
Inclusion Criteria:

* age: 18- 80
* diagnosis of psoriasis vulgaris (mild- middle)
* no other current antipsoriatic therapy (systemic/topical)
* at least 5 psoriatic areas of 5x5 cm

Exclusion Criteria:

* pregnancy/nursing mothers
* women in reproductive age without adequate contraception
* severe and acute forms of psoriasis vulgaris
* patients receiving systemic or topical antipsoroatic treatment in past 3 month
* UV-therapy in past 3 month
* patients having a positive anamnesis for squamous cell carcinoma, malignant melanoma, basalioma
* epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
PASI, PGA | 4 weeks

SECONDARY OUTCOMES:
OCT/ultrasound- thickness of epidermis/ dermis | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Wozel, Prof. Dr.med, Principal Investigator — Department of Dermatology, Medical Faculty, Technical University Dresden, Germany
Locations (1):
- Department of Dermatology, Medical Faculty, TU Dresden, Dresden, Germany